CLINICAL TRIAL: NCT04127344
Title: Effect of a Music Therapy Intervention on the Mood of the Critical Patient in a Tertiary Hospital.
Brief Title: Effect of a Music Therapy Intervention on Mood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-MUS-2018-83
Record Dates: First submitted 2019-08-29; First posted 2019-10-15 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Critically Ill Patient

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, parallel and open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy Intervention (Experimental): Patients enrolled will be randomised between two arms: Music Therapy Intervention and Non-Music Therapy Intervention.
  Patients randomised to a music therapy intervention will receive an individualised music therapy intervention.
  Interventions: Behavioral: Music Therapy Intervention
- Non-Music Therapy Intervention (No Intervention): Patients enrolled will be randomised between two arms: Music Therapy Intervention and Non-Music Therapy Intervention.
  Patients allocated to Non-Music Therapy Intervention received standard treatment.

INTERVENTIONS:
Behavioral: Music Therapy Intervention — Patients randomized to a music therapy intervention will receive an individualised music therapy intervention. The sessions will last 10-20 minutes and they will be done by music therapist and musician.
  Arms: Music Therapy Intervention

SUMMARY:
The hypothesis is that the music therapy intervention has a positive impact on the critical patients' mood as it has a reassuring effect that allows a connection with emotions, helps to communicate and affects the welfare of patients. It also reduces pain and the consumption of painkillers and sedatives, as well as vasoactive drugs in critical patients.

DETAILED DESCRIPTION:
The aim of the study is to assess the effect of a personalised music therapy intervention with standard treatment on critical patients' mood compared to those who just receive the standard treatment. Moreover, the effect of the different interventions on pain and sedative, analgesic and vasoactive drugs will also be assessed.

This is a randomized, parallel and open clinical trial that will compare: a) a music therapy intervention combined with the standard care (experimental group), with b) standard care (control group), on critical patients admitted to the General, Cardiac and Coronary Intensive Care Unit of the Santa Creu I Sant Pau Hospital.

The expected number of patients expected to be included in this trial is 164. Patients will be included and randomized the day the music therapy intervention is to take place, once a week. Patients' mood will be assessed with a validated questionnaire in Spanish for adults, the POMS (Profile of Mood States) survey that consists of a self-report built on the basis of a multidimensional conception of mood and has a Likert 5-points type format (0 to 4)

ELIGIBILITY:
Inclusion Criteria:

* Patients who are oriented in time, space and person
* Glasgow Coma Scale of 15 or 11+intubated
* Negative the Confusion Assessment Method for the ICU (CAM-ICU)
* Richmond Agitation-Sedation Scale of 0
* Patients who are at least conscious and oriented for 48 hours in the ICU.

Exclusion Criteria:

* Auditory deficit
* Patients that have participated in the study previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-03-12 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mood state | 24 hours
  The mood state will be assessed through the Profile of Mood States Scale (POMS) after randomization, within the next 6 to 12 hours, and 24 hours after randomization.

SECONDARY OUTCOMES:
Level of pain | 24 hours
  The level of pain will be assessed through an Analogical Visual Scale after randomization, within the next 6 to 12 hours, and 24 hours after randomization.
Consumption of analgesics and sedatives | 24 hours
  Consumption of analgesics and sedatives will be assessed after randomization, within the next 6 to 12 hours, and 24 hours after randomization.
Consumption of vasoactive drugs | 24 hours
  Consumption of vasoactive drugs will be assessed after randomization, within the next 6 to 12 hours, and 24 hours after randomization.
Physiological variables (blood pressure, heart rate, breathing rate and oxygen saturation) | 24 hours
  The physiological variables will be assessed after randomization, within the next 6 to 12 hours, and 24 hours after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Mª del Mar Vega Castosa, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain